CLINICAL TRIAL: NCT05212181
Title: Smart Robot Therapy for Stroke Upper Limb Rehabilitation: A Proof-of-value Trial of Clinic to Home Robotics-assisted Telerehabilitation
Brief Title: Clinic to Home Robotics-assisted Telerehabilitation for Upper Limb (CHISEL)
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: ARTICARES Pte Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: DSRB 2021/00156
Record Dates: First submitted 2022-01-18; First posted 2022-01-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: H-Man — H-Man device will be deployed to patients for onboarding and home-based training.

SUMMARY:
Hemiparetic weakness is common after stroke and only a small group of patients achieve useful upper limb function despite best rehabilitation efforts. This is due to the lack of intensive upper limb therapies to drive neuroplasticity either in clinic or at home.

In this study, we plan to pilot home-based, robot-aided-therapy using H-man to deliver intensive arm rehabilitation.

DETAILED DESCRIPTION:
It has been assumed that stroke survivors reach a plateau in their recovery within 3-6 months of their stroke. They tend to receive minimal rehabilitation support once they are discharged to the community citing obstacles such as ambulation, transportation, and cost.

H-man is a novel telerehabilitation, upper limb training robot, that will deliver robot-aided therapy in patients' homes by clinic-based therapists through remote monitoring and under the supervision of their caregivers.

The study aims to refine and evaluate the feasibility, efficacy and safety of home-based training using the H-man robot.

ELIGIBILITY:
Inclusion Criteria:

1) Clinical stroke (ischaemic or haemorrhagic) confirmed by admitting doctors and CT, CT angiography or MRI brain imaging (2) Age 21 to 90 years, both males and females (3) At least > 28 days (4) Upper limb motor impairment of Fugl-Myer Motor Assessment (FMA) scale 10 to 60 (5) Has a stable home abode and a carer/ NOK to supervise home based exercise. (6) Ability to sit supported continuously for 60 minutes (7) Montreal Cognitive Assessment (MOCA) score > 21/30 (8) Able to understand purpose of research and give consent

Exclusion Criteria:

1. Non-stroke related causes of arm motor impairment
2. Medical conditions incompatible with research participation: uncontrolled medical illnesses (hypertension or diabetes, ischaemic heart disease, congestive heart failure, bronchial asthma, severe /untreated depression, agitation, end stage renal/liver/heart/lung failure, unresolved cancers.
3. Anticipated life expectancy of < 6 months
4. Inability to tolerate sitting continuously for 60 minutes (5 Local factors potentially worsened by intensive robot-aided arm therapy and computer-based training: active seizures within 3 months, spasticity of Modified Ashworth Scale grades >2 skin wounds, shoulder, arm pain VAS >5/10, active upper limb fractures, arthritis, fixed upper limb flexion contractures.

(6) Hemi anaesthesia of affected limb (7) Severe visual impairment or visual neglect affecting ability to use H-Man robot (8) History of dementia, severe depression or behavioural problems (9) Pregnant or lactating females will not be allowed to participate (10) Absence of reliable carer to provide supervision during home training.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Motor Assessment | Assessed at week 5 from baseline (week 0)
  Change in Fugl Meyer Motor Assessment score in the affected arm

SECONDARY OUTCOMES:
Aggregated number | Assessed at weeks 0, 5, 12 and 24
  Mean/day and total cumulative over 30 days H-Man robot recorded arm repetitions (robotic metrics)
Streamlined Wolf-motor function test (SWMFT) | Assessed at weeks 0, 5, 12 and 24
  Functional score for stroke patients, minimum 0, maximum 75; with higher score indicating better function
Action Research Arm Test (ARAT) | Assessed at weeks 0, 5, 12 and 24
  Functional and dexterity score for upper extremities, minimum 0, maximum 57; with higher score indicating better function
Grip strength (KgF) measured by Digital Dynamometer (mean of 3 readings will be recorded) | Assessed at weeks 0, 5, 12 and 24
  Measured by Digital Dynamometer (mean of 3 readings will be recorded)
Self-efficacy outcomes by UPSET (upper limb self-efficacy test) | Assessed at weeks 0, 5, 12 and 24
  Questionnaire to measure self-efficacy in various tasks after stroke
HrQOL scales using SS-QOL (Stroke specific Quality of Life scale) | Assessed at weeks 0, 5, 12 and 24
  Quality of life scale specific to stroke patients, minimum 49, maximum 245; with higher scores indicating better function
PROMs using subjective scales (Likert 0-5) to questions | Assessed at weeks 0, 5, 12 and 24
  E.g. how beneficial, how comfortable, how useful, how easy was H-Man robot training experience at home, and would they prefer this to be part of standard therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Poo Lee Ong, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aguirre-Ollinger G, Chua KSG, Ong PL, Kuah CWK, Plunkett TK, Ng CY, Khin LW, Goh KH, Chong WB, Low JAM, Mushtaq M, Samkharadze T, Kager S, Cheng HJ, Hussain A. Telerehabilitation using a 2-D planar arm rehabilitation robot for hemiparetic stroke: a feasibility study of clinic-to-home exergaming therapy. J Neuroeng Rehabil. 2024 Nov 26;21(1):207. doi: 10.1186/s12984-024-01496-6. PMID 39593101